CLINICAL TRIAL: NCT02355483
Title: Accuracy of Unenhanced CT in Elderly Patients Admitted to the Emergency Department With Acute Abdominal Symptoms
Brief Title: Impact of Unenhanced Computed Tomography (CT) in Elderly Patients Admitted to the Emergency Department With Acute Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8741; 2011-A00868-33 (Other: AFSSAPS)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Unenhanced abdominal Computed Tomography — Systematic Unenhanced abdominal Computed tomography

SUMMARY:
The purpose of this study is to determine whether non-contrast abdominal computed tomography (CT) impacts management (diagnosis, need for surgery and treatment) in elderly patients admitted to the emergency department with abdominal pain.

DETAILED DESCRIPTION:
A systematic unenhanced abdominal CT is performed in elderly patients admitted to the emergency patients with acute abdominal symptoms. Accuracy of unenhanced CT is assessed by comparing diagnosis and therapeutic management recorded before and after unenhanced CT versus gold standard diagnosis and management. Gold standard diagnosis and management are established at 3 month follow up, based on patient's medical records and a systematic telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients admitted to the emergency department (aged 75 year old and older)
* acute abdominal pain
* informed consent

Exclusion criteria:

* traumatic pain
* symptom duration of more than a week
* unability for the patient to give informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 423 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 3 months
  Emergency Department (ED) diagnosis made prospectively by the attending ED physician both before and after unenhanced abdominal CT is compared to the reference diagnosis established at 3 month follow-up. Both ED diagnosis and reference diagnosis are recorded using a standardized diagnosis list.

SECONDARY OUTCOMES:
Therapeutic management accuracy | 3 months
  Therapeutic management made by the attending ED physician both before and after unenhanced abdominal CT is compared to reference management established at 3 month follow-up. Therapeutic management is assessed by patient orientation following ED admission, need for hospitalization and surgical or medical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid MILLET, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Medical Imaging department, Montpellier, France